CLINICAL TRIAL: NCT01558570
Title: Intracellular Tight Junction Permeability in Schizophrenia: Focus on Zonulin
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University of Maryland, College Park (Other)
Responsible Party: Principal Investigator, MPRC, Deanna L. Kelly, Pharm.D., BCPP, University of Maryland, Baltimore
Other Study IDs: HP-00049310
Record Dates: First submitted 2011-09-12; First posted 2012-03-20 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Schizophrenia; Celiac Disease
MeSH Terms: conditions — Schizophrenia; Celiac Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Laboratory Measures:
  Zonulin and gliadin antibodies will be sent to the lab of Dr. Alessio Fasano for assay.
  Genetic and Biochemical analysis will be sent for analysis and storage of blood sample at the Maryland Psychiatric Research Center Neurogenetics laboratory under the direction of Dr. Ikwunga Wonodi. Analysis will include kynurenic acid metabolites, inflammatory markers from Peripheral Blood Mononuclear Cells (PBMC) and future genetic analysis including but not limited to human leukocyte antigen (HLA) haplotypes (DQ2 and DQ8).
  Cytokines will be analyzed by the Cytokine Core Laboratory at the University of Maryland using Luminex Technology.
  Other standard laboratories will be done by Lab Corp or other contract laboratory.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Schizophrenia
  Interventions: Procedure: Blood Draw

INTERVENTIONS:
Procedure: Blood Draw — One time blood draw

SUMMARY:
The purpose of this protocol is to collect serum zonulin levels in people with schizophrenia. This one time visit will collect zonulin levels, antibodies to gliadin (tissue transglutaminase and antigliadin antibodies) and other information that may relate to increased intracellular tight junction permeability as it related to the immune and stress system and the immune association with kynurenic acid pathway 50. Data will be collected for use in future grant applications and published reports.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV Diagnosis of Schizophrenia or Schizoaffective Disorder
* Male or females between ages of 18 to 75 years

Exclusion Criteria:

* Score below 10/12 on the Evaluation to Sign Consent (ESC)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with schizophrenia will be recruited by MPRC through their patient recruiting network including the Treatment Research Program and the Outpatient Research Program and affiliated sites. Patient with schizophrenia may also be recruited through the NIDA screening protocol process. (UMB approved IRB protocol HP-00043664)
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Zonulin concentration in serum (ng/mg) | 1 day
  Participants will undergo a one-time blood draw in order to test for zonulin concentration in serum (ng/mg) and these results will be compared to normative data to screen for elevations. The sample size for this pilot study was estimated based on the known prevalence of Celiac disease in schizophrenia, a disease known to have elevated zonulin levels.

CONTACTS AND LOCATIONS:
Overall Officials: Deanna L. Kelly, Pharm.D., BCPP, Principal Investigator — University of Maryland, College Park
Locations (1):
- Maryland Psychiatric Research Center, Catonsville, Maryland, United States

REFERENCES:
- See also: Maryland Psychiatric Research Center — http://www.mprc.umaryland.edu